CLINICAL TRIAL: NCT02776527
Title: A Clinical Trial of Maintenance Treatment of Apatinib in Advanced Gastric Cancer Patients Have Completed Postoprative Adjuvant Chemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBG001
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; D2 Lymphadenectomy; postoprative adjuvant chemotherapy; Apatinib; disease free survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A group (Experimental): D2 Radical Gastrectomy adding received postoprative adjuvant chemotherapy of eight cycles of Xelox,and taking Apatinib 500mg/qd orally, 28 days as a cycle, till disease progresses.
  Interventions: Drug: Apatinib Mesylate Tablets
- B group (No Intervention): D2 Radical Gastrectomy adding received postoprative adjuvant chemotherapy of eight cycles of Xelox

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — taking Apatinib Mesylate Tablets 500mg/qd orally, 28 days as a cycle, till disease progresses
  Other Names: AiTan
  Arms: A group

SUMMARY:
The main purpose of this study is to evaluate whether the Apatinib can improve the disease free survival (DFS) of gastric cancer patients in stage IIIB/IIIc, who had completed postoprative adjuvant chemotherapy. Meanwhile, the investigators also will evaluate whether the Apatinib can improve the overall survival (OS), estimate the quality of life of patients have taken the Apatinib and monitor the security of Apatinib.

DETAILED DESCRIPTION:
The investigators will recruit 40 gastric cancer patients who underwent D2 lymphadenectomy and histologically verified as stage ⅢB or ⅢC according to the seventh edition of the TNM classification for gastric cancer. When these patients have completed 8 cycles of Xelox as adjuvant chemotherapy without any recurrence, they will randomly assigned to group A or B. Each group possesses 20 gastric cancer patients finally. Patients in group A will receive the best supportive care，and take Apatinib 500mg/qd orally, 28 days as a cycle, till disease progresses. Patients in group B will receive the best supportive care. Through follow-up and statistics, the investigators will observe whether Apatinib can improve the disease free survival (DFS) of gastric cancer patients with stage IIIb&IIIC. Meanwhile, the investigators also will observe whether the Apatinib can improve the overall survival (OS) and estimate the quality of life of patients have taken the Apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients ranges from 18 to75 years old.
2. Score of the Eastern Cooperative Oncology Group (ECOG) performance status ranges from 0 to 2.
3. All tumor tissues were histologically verified as advanced gastric cancer, and patients with no less than 15 dissected lymph nodes and stage of ⅢB or ⅢC according to TNM, were chosen.
4. Gastric cancer patients underwent the curative gastrectomy with D2 lymphadenectomy.
5. Gastric cancer patients received postoprative adjuvant chemotherapy of eight cycles of Xelox. During the period of chemotherapy, no one relapses. If the patients could well tolerate the adjuvant chemotherapy, it is recommended that patients can obtain maintenance treatment of Apatinib after postoprative adjuvant chemotherapy of eight cycles of Xelox.
6. Previously, patients did not receive the therapy of Apatinib or other VEGFR inhibitor, such as Sorafenib, Sunitinib.
7. The blood examination is normal: neutrophil count≥1.5×109/L；hemoglobin≥80 g/L；blood platelet count≥100×109/L；total bilirubin≤1.5×ULN；ALT、AST≤2.5×ULN；
8. Patients have no serious heart, lung, liver, kidney diseases and jaundice and digestive tract obstruction. Patients have no an acute infection.

   -

Exclusion Criteria:

1. The score of KPS<60 or anticipated survival time<3 months.
2. Previously, patients received neoadjuvant chemotherapy.
3. Within six months, patients encountered heart cerebral disease, got an uncontrolled hypertension (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg), had serious coronary heart disease, serious arrhythmia, first-grade cardiac insufficiency. Patients have positive urinary protein.
4. Patients have clear gastrointestinal bleeding tendency, local active ulcer lesions, fecal occult blood (++); Patients have the symptoms of melena and haematemesis within 2 months.
5. Coagulopathy (INR>1.5、APTT>1.5 ULN), hemorrhage tendency.
6. Patients have these symptoms, such as dysphagia, nausea, vomiting, chronic diarrhea and intestinal obstruction.
7. Patients have these symptoms, such as neurological diseases, mental illness, serious infection.
8. Patients were pregnant, in nursing, or have bearing requirement during the study period.
9. Patients got other primary malignant tumors (except curable skin basal cell carcinoma and cervical cancer in situ) except gastric cancer within 5 years.
10. Patients have distant metastasis.
11. Within 6 months before study starts and in the process of this study, patients participate in other clinical researches.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 2 years
  Disease free survival (DFS) was defined as the length of time from the date of randomization to the date of first documentation of relapse of gastric cancer or any other type of cancer or death.

SECONDARY OUTCOMES:
overall survival | 3 years
  Overall survival (OS) was defined as the length of time from the date of randomization to the date of death of various reasons

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, Master, Principal Investigator — Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China